CLINICAL TRIAL: NCT00760383
Title: Muscle Regrowth During Physical Rehabilitation and Amino Acid Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Hans Dreyer, University of Oregon, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1K01HD057332 (NIH); 1K01HD057332 (NIH)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis
Keywords: Total Knee Arthroplasty; Osteoarthritis; Muscle Metabolism; Rehabilitation; Physical Therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Amino Acids, Essential; Histidine; Isoleucine; Leucine; Lysine; Methionine; Phenylalanine; Threonine; Valine; Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EAA+PT (Experimental): 20 g EAA daily for 7 days prior to TKA surgery and for 14 days after surgery.
  Interventions: Dietary Supplement: Essential amino acids
- ALA+PT (Placebo Comparator): 20 g NEAA daily for 7 days prior to TKA surgery and for 14 days after surgery.
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Essential amino acids — Subjects will ingest 20 grams of essential amino acids (EAA) daily for 7 days prior to total knee arthroplasty (TKA) surgery and for 14 days after surgery daily. On the days they are seen by physical therapy (PT) they will ingest the EAA supplement 30 minutes after the end of each PT rehabilitation session.
  Other Names: Histidine; Isoleucine; Leucine; Lysine; Methionine; Phenylalanine; Threonine; Valine
  Arms: EAA+PT
Dietary Supplement: Alanine — Subjects will ingest 20 grams of non-essential amino acid (NEAA) daily for 7 days prior to total knee arthroplasty (TKA) surgery and for 14 days after surgery daily. On the days they are seen by physical therapy (PT) they will ingest the NEAA supplement 30 minutes after the end of each PT rehabilitation session.
  Arms: ALA+PT

SUMMARY:
The general hypothesis is that in older adults muscle regrowth after an acute musculoskeletal stress will be positively influenced by traditional physical rehabilitation, and further enhanced by nutritional supplementation. Using state-of-the-art stable isotope methodologies for the study of muscle metabolism and methodologies for the measurement of cell signaling, we will test the following specific hypotheses: 1) Total knee arthroplasty (TKA) induces an acute net protein catabolism mainly by reducing muscle protein synthesis; 2) TKA induced catabolism is attenuated by the ingestion of essential amino acids (EAA); 3) EAA supplementation in combination with physical therapy (PT) will stimulate muscle protein synthesis and mTOR signaling to a greater extent than PT with Placebo; and 4) EAA supplementation during TKA PT rehabilitation will improve muscle strength, muscle volume and functional outcomes to a greater extent than PT with Placebo.

Public Benefit: This research will focus rehabilitation efforts on specific and currently unresolved mechanisms responsible for muscle loss following total knee replacement in older adults. While knee pain due to bone arthritis is often alleviated after knee replacement, complete return of physical function and independence is difficult to achieve. This research will help to restore physical function and independence in the rapidly growing population of older adults with knee arthritis.

DETAILED DESCRIPTION:
The goal of this translational research project is to identify key mechanisms involved in regulating skeletal muscle loss and regrowth following total knee arthroplasty (TKA). Total knee arthroplasty induces significant declines in muscle mass and strength, which is directly responsible for reduced function, specifically functional independence. Such declines in muscle strength and volume and activities of daily living (getting up from a chair, climbing stairs and walking) can persist for up to 2 years.

Atrophy is the direct result of an imbalance between muscle protein synthesis and breakdown. However, there are two quite distinct mechanisms leading to muscle loss: accelerated protein breakdown (e.g. burn injury), primarily resulting from the stress response, or decreased protein synthesis (e.g., immobilization). In case of severe stress, muscle protein synthesis actually increases, although not adequately to impede muscle loss, and anabolic stimuli, such as nutrition, cannot counteract muscle atrophy. On the other hand, decreased protein synthesis from inactivity can be stimulated by nutrition and exercise, thereby reducing or preventing atrophy. Currently, we do not know which condition predominates following TKA: surgical stress-induced catabolism or immobility-associated declines in synthesis . What is not known is which signaling pathway predominates following TKA; stress induced catabolism or immobility associated declines in synthesis. Our goal is to determine which model (stress or inactivity) accounts for the acute and rapid muscle loss following TKA in order to better focus rehabilitation efforts.

Our general hypothesis is that quadriceps atrophy following TKA surgery is primarily due to inactivity, which can be counteracted by physical therapy (PT) and essential amino acid (EAA) supplementation. Our goal is to delineate the basic mechanisms underlying muscle loss with TKA, and based on this new information, to find novel rehabilitation strategies to accelerate recovery of normal function from TKA.

Thus, our plan is to test in older adults the following specific hypothesis:

1. TKA induces an acute and severe net protein catabolism by reducing muscle protein synthesis
2. TKA induced catabolism is attenuated with the ingestion of EAA
3. EAA supplementation following PT will stimulate muscle protein synthesis and mTOR signaling to a greater extent than PT with Placebo
4. EAA supplementation during TKA PT rehabilitation will improve muscle strength, muscle volume and functional outcomes to a greater extent than PT with Placebo

To test our specific hypothesis we will address the following specific aims:

1. To determine if TKA surgery reduces muscle protein synthesis and/or increases muscle protein breakdown
2. To determine if muscle protein synthesis is acutely increased with the ingestion of EAA following TKA surgery
3. To determine if muscle protein synthesis and mTOR signaling will be stimulated by PT rehabilitation and enhanced by EAA supplementation
4. To determine if EAA supplementation during TKA with traditional PT for 6 weeks improves muscle strength, muscle volume and functional outcomes This application will provide preliminary data for the submission of an R01 grant to further determine the mechanisms leading to successful return of quadriceps muscle strength and function following TKA. Essential amino acids are inexpensive, well tolerated and easily digestible and have been shown to independently stimulate muscle protein synthesis and components of the anabolic mTOR signaling pathway. My goal of increasing muscle strength and functional mobility is specifically outlined in the National Center for Medical Rehabilitation Research Seven Priority Areas and are in line with the NIH roadmap and priorities, and will help us to understand muscle protein metabolism during physical therapy rehabilitation. By adopting a mechanism-driven, translational research design that links changes in cell signaling with functional outcome measures (cell → system → function) we will capture key physiological events responsible for the regulation of muscle mass and function following TKA.

ELIGIBILITY:
Inclusion Criteria:

* Total Knee Arthroplasty surgical candidate

Exclusion Criteria:

* Overt muscle disease

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Dreyer, PT, PhD, Principal Investigator — Assistant Professor, Department of Human Physiology
Locations (2):
- United States (2):
  - University of Oregon, Eugene, Oregon
  - Slocum Center for Orthopedics and Sports Medicine, Eugene, Oregon

REFERENCES:
- [Background] Dreyer HC, Drummond MJ, Pennings B, Fujita S, Glynn EL, Chinkes DL, Dhanani S, Volpi E, Rasmussen BB. Leucine-enriched essential amino acid and carbohydrate ingestion following resistance exercise enhances mTOR signaling and protein synthesis in human muscle. Am J Physiol Endocrinol Metab. 2008 Feb;294(2):E392-400. doi: 10.1152/ajpendo.00582.2007. Epub 2007 Dec 4. PMID 18056791
- [Background] Fujita S, Dreyer HC, Drummond MJ, Glynn EL, Cadenas JG, Yoshizawa F, Volpi E, Rasmussen BB. Nutrient signalling in the regulation of human muscle protein synthesis. J Physiol. 2007 Jul 15;582(Pt 2):813-23. doi: 10.1113/jphysiol.2007.134593. Epub 2007 May 3. PMID 17478528
- [Background] Dreyer HC, Fujita S, Cadenas JG, Chinkes DL, Volpi E, Rasmussen BB. Resistance exercise increases AMPK activity and reduces 4E-BP1 phosphorylation and protein synthesis in human skeletal muscle. J Physiol. 2006 Oct 15;576(Pt 2):613-24. doi: 10.1113/jphysiol.2006.113175. Epub 2006 Jul 27. PMID 16873412
- [Background] Fujita S, Dreyer HC, Drummond MJ, Glynn EL, Volpi E, Rasmussen BB. Essential amino acid and carbohydrate ingestion before resistance exercise does not enhance postexercise muscle protein synthesis. J Appl Physiol (1985). 2009 May;106(5):1730-9. doi: 10.1152/japplphysiol.90395.2008. Epub 2008 Jun 5. PMID 18535123
- [Background] Drummond MJ, Dreyer HC, Pennings B, Fry CS, Dhanani S, Dillon EL, Sheffield-Moore M, Volpi E, Rasmussen BB. Skeletal muscle protein anabolic response to resistance exercise and essential amino acids is delayed with aging. J Appl Physiol (1985). 2008 May;104(5):1452-61. doi: 10.1152/japplphysiol.00021.2008. Epub 2008 Mar 6. PMID 18323467
- [Background] Dreyer HC, Blanco CE, Sattler FR, Schroeder ET, Wiswell RA. Satellite cell numbers in young and older men 24 hours after eccentric exercise. Muscle Nerve. 2006 Feb;33(2):242-53. doi: 10.1002/mus.20461. PMID 16315322
- [Background] Dreyer HC, Volpi E. Role of protein and amino acids in the pathophysiology and treatment of sarcopenia. J Am Coll Nutr. 2005 Apr;24(2):140S-145S. doi: 10.1080/07315724.2005.10719455. PMID 15798081
- [Result] Ratchford SM, Bailey AN, Senesac HA, Hocker AD, Smolkowski K, Lantz BA, Jewett BA, Gilbert JS, Dreyer HC. Proteins regulating cap-dependent translation are downregulated during total knee arthroplasty. Am J Physiol Regul Integr Comp Physiol. 2012 Mar 15;302(6):R702-11. doi: 10.1152/ajpregu.00601.2011. Epub 2011 Dec 28. PMID 22204954
- [Derived] Dreyer HC, Strycker LA, Senesac HA, Hocker AD, Smolkowski K, Shah SN, Jewett BA. Essential amino acid supplementation in patients following total knee arthroplasty. J Clin Invest. 2013 Nov;123(11):4654-66. doi: 10.1172/JCI70160. Epub 2013 Oct 25. PMID 24135139
- See also: Clinical and translational research on skeletal muscle physiology before, during and after total knee arthroplasty (TKA) surgery — http://muscle.uoregon.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Slocum Center for Orthopedics and Sports Medicine.
Pre-assignment Details: Participants were selected from surgical candidates from the Slocum Center for Orthopedics and Sports Medicine. All subjects were scheduled to undergo primary TKA.
Period: Overall Study
Arm/Group | EAA+PT | ALA+PT
Started | 21 | 19
Completed | 16 | 12
Not Completed | 5 | 7
Not completed — moved away; withdrew; medical reasons | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EAA+PT | ALA+PT | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (5) | 70 (5) | 69 (5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 15 | 17 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Stair Time up
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | EAA+PT | ALA+PT
Number analyzed (Participants) | 16 | 12
seconds | 7 (1) | 8 (1)

2. Primary Outcome: Quadriceps Muscle Strength
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: Newtons
Arm/Group | EAA+PT | ALA+PT
Number analyzed (Participants) | 16 | 12
Newtons | 65 (8) | 81 (7)

3. Secondary Outcome: Mid-thigh Muscle Volume
Description: Analysis was performed using the Analyze 11 software package with semi-automated delineation of quadriceps, hamstrings, and adductors boarders. Using thresholding methods, the software can differentiate operator-delineated parameters set to distinguish muscle from non-muscle (i.e., adipose tissue) using voxel intensity within each border region for quantitative determination of muscle volume.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: Volume (cm^3)
Arm/Group | EAA+PT | ALA+PT
Number analyzed (Participants) | 16 | 12
Volume (cm^3) | 109 (11) | 108 (9)

ADVERSE EVENTS:
Arm/Group | EAA+PT | ALA+PT
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No